CLINICAL TRIAL: NCT04734574
Title: Use of Different Methods of Confirmation of Brain Death in Brain Death Donors
Brief Title: Methods of Confirmation of Brain Death
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Ondrej Hrdy, Principal Investigator, Brno University Hospital
Other Study IDs: CT0022020
Record Dates: First submitted 2021-01-26; First posted 2021-02-02 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Brain Death; Organ Donation
MeSH Terms: conditions — Brain Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to describe the use of methods confirming brain death in the real clinical practice of the transplant program in the Czech Republic.

DETAILED DESCRIPTION:
Organ donation is possible in the Czech Republic only after meeting the legislative requirements. These require confirmation of brain death by one of the statutory methods before organ harvesting. The use of these methods in clinical practice has not yet been described.The aim of this retrospective observational study is to describe the use of these methods in the real clinical practice of the transplant program in the Czech Republic, taking into account the legislation of other European countries.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* organ donor

Exclusion Criteria:

* age under 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult critically ill patinets with confirmed brain death admitted to university hospital who become brain death organ donor.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Angiography | within 24 hours after the onset of signs of brain death
  Cerebral panangiography
Brainstem auditory evoked potentials | within 24 hours after the onset of signs of brain death
  Brainstem auditory evoked potentials
Brain scintigraphy | within 24 hours after the onset of signs of brain death
  Brain scintigraphy
Cerebral computed tomography angiography | within 24 hours after the onset of signs of brain death
  Cerebral computed tomography angiography
Transcranial Doppler ultrasonography | within 24 hours after the onset of signs of brain death
  Transcranial Doppler ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Roman Gal, M.D., Ph.D., Study Chair — University Hospital Brno
Locations (1):
- University Hospital Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No